CLINICAL TRIAL: NCT02243436
Title: Phase I-II Clinical Trial for the Evaluation of Brentuximab Vedotin Plus Etoposide, Solumoderin (Methylprednisolone), High Dose ARA-C (Cytarabine) and Cisplatin in the Transplant and Post-transplant Management for Relapsed or Refractory Classical Hodgkin Lymphoma Patients
Brief Title: Brentuximab Vedotin in Pre-transplant Induction and Consolidation for Relapsed or Refractory Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Grupo Español de Linfomas y Transplante Autólogo de Médula Ósea (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRESHAP-GELTAMO.LH-2013; 2014-000835-17 (EudraCT Number)
Record Dates: First submitted 2014-08-27; First posted 2014-09-18 (Estimated); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: CLASSICAL HODGKIN LYMPHOMA
Keywords: CLASSICAL HODGKIN LYMPHOMA; HODGKIN LYMPHOMA; LYMPHOMA; HL
MeSH Terms: conditions — Hodgkin Disease; Lymphoma | interventions — Brentuximab Vedotin; Etoposide; Methylprednisolone; Cisplatin; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BV-ESHAP (Experimental): 1. - 3 cycles every 21 days:
     * Brentuximab Vedotin, on day 1 (BV will be administered at three different doses 0.9mg/kg, 1.2mg/kg, 1.8mg/kg)
     * Etoposide 40 mg/m2/day, on days 1 to 4
     * Soludomerin (methylprednisolone) 250 mg/day, on days 1 to 4
     * Cisplatin 25 mg/m2/day, on days 1 to 4
     * Ara C (cytarabine) 2 g/m2, on day 5
  2. - A fourth dose of BV will be given 21 days after the third BV dose during the evaluation of response before the transplant.
  3. - Autologous peripheral blood stem cell transplant
  4. - A fifth dose of BV (1.8mg/kg) will be given on between day 28 and 35 post-transplant, followed by two additional doses (1.8mg/kg) every 3 weeks, to complete a total of 7 BV infusions.
  Interventions: Drug: Brentuximab Vedotin; Drug: Etoposide; Drug: Soludomerin; Drug: Cisplatin; Drug: Ara C

INTERVENTIONS:
Drug: Brentuximab Vedotin — Brentuximab Vedotin, 0.9mg/kg, 1.2mg/kg, 1.8mg/kg, day 1
  Other Names: ADCETRIS
Drug: Etoposide — Intravenose use, 40mg/m2/day, on days 1 to 4
Drug: Soludomerin — Intravenous use, 250mg/day, on days 1 to 4
  Other Names: Methylprednisolone
Drug: Cisplatin — Intravenous use, 25mg/m2/day, on days 1 to 4
Drug: Ara C — Intravenous use, 2g/m2, day 5
  Other Names: Cytarabine

SUMMARY:
Phase I trial aimed to determine the Maximum Tolerable Dose of the BV in combination with ESHAP in relapsed/resistant Hodgkin Lymphona patients and to evaluate response to treatment with BV-ESHAP as salvage regimen prior to autologous stem cell transplantation.

DETAILED DESCRIPTION:
Most patients suffering from Hodgkin's lymphoma (HL) can be successfully treated with standard chemo- and/or radiotherapy. However, in patients with refractory disease/relapsing after first line of therapy, conventional-dose chemotherapy regimens induce low remission rates, with long-term disease free survival not higher than 10% of patients.

High-dose chemotherapy followed by autologous stem cell transplantation (ASCT) has become the standard treatment for these patients. This treatment approach results in long-term remissions in approximately 40-50% of relapsed patients, and in up to 25-30% of those with primary refractory disease. The possibility of a cure depends on several prognostic factors, however, in almost all series, the strongest prognostic factor has been the disease status before ASCT. Patients with HL who do not achieve complete remission (CR) after induction chemotherapy and those with unresponsive relapse have a very poor prognosis. Therefore, the choice of a very active pre-transplant salvage chemotherapy regimen is extremely important to improve results after ASCT. In addition, this activity should also be combined with a good stem cell mobilizing potential and low toxicity profiled.

Several pre-transplant salvage regimens for refractory/relapsed HL are currently used with an overall response (OR) and CR rates ranging from 60% to 88% and from 17% to 49%, respectively. No randomized trial exists comparing the effectiveness of these regimens. ESHAP (Etoposide, Solumoderin (methylprednisolone), Ara-C (Cytarabine) and cisplatin) is one of the most commonly used regimens. ESHAP induces an OR and CR of 73% and 41%, respectively, with 5% toxic deaths. In the present study, a combination of ESHAP plus Brentuximab Vedotin (BV) is proposed as pre-transplant therapy with the aim to improve the CR rate before ASCT.

HL is characterized by the presence of CD30-positive Hodgkin Reed-Sternberg cells. The antibody-drug conjugate BV delivers the highly potent antimicrotubule agent monomethyl auristatin E (MMAE) to CD30-positive malignant cells by binding specifically to CD30 on the cell surface and releasing MMAE inside the cell via lysosomal degradation.

Binding of MMAE to tubulin results in apoptotic death of the CD30 expressing tumor cell.

ELIGIBILITY:
Inclusion Criteria:

Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study

* Histologically confirmed relapsed or refractory classical HL after first line chemotherapy. CD30 has to be positive
* Age 18 to 65 years. Patient >65 years old with ECOG ≤1 and absence of comorbidities will be included in the study
* ECOG ≤2
* Karnofsky performance status ≥ 60
* No major organ dysfunction
* Biopsy at HL relapse or when refractoriness disease is diagnosed must be done prior to BV-ESHAP. If biopsy cannot be performed, tumor biopsy at initial diagnosis of HL must be available to be revised
* Absence of prior history of other malignant diseases, except:

Basal cell carcinoma of the skin or uterine "in situ" carcinoma adequately treated Any curable neoplasia adequately treated that has achieved complete response and has remained in such status longer than 3 years

* Female patient is either post-menopausal for at least 1 year before the screening visit or surgically sterile or if of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 30 days after the last dose of study drug, or agrees to completely abstain from heterosexual intercourse
* Male patients, even if surgically sterilized, agree to practice effective barrier contraception during the entire study period and through 6 months after the last dose of study drug, or agrees to completely abstain from heterosexual intercourse
* Life-expectancy >3 months
* Platelet count ≥75•109/L (or 20 if due to Bone Marrow [BM] infiltration) absolute neutrophil count ≥1.5•109/L (or 0.5 if due to BM infiltration), and hemoglobin ≥ 8g/dL
* Total Bilirubin: <1.5 x UNL, unless clearly related to the disease (Gilbert disease will be ruled out from this point)
* AST and ALT: <3 xUNL except liver infiltration
* Serum creatinine: < 2.0 mg/dL and/or creatinine clearance or calculated creatinine clearance > 40 mL/minute
* Serum sodium >130 mmol/L
* Voluntary written informed consent

Exclusion Criteria:

* Current active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases or stable chronic liver disease per investigator assessment)
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Patients that have been treated previously with anti-CD30 monoclonal antibodies
* Myocardial infarction within 6 months prior to enrollment. Heart failure NYHA Class III-IV, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Recent evidence (within 6 months) of a left-ventricular ejection fraction <50%
* Peripheral neuropathy or neuropathic pain grade ≥ 2
* Known cerebral or meningeal disease, including signs or symptoms of PML
* Symptomatic neurologic disease compromising normal activities of daily living or requiring medication
* Known hypersensitivity to recombinant proteins, murine proteins, or to any excipient contained in brentuximab vedotin
* Pregnant women or in breast-feeding period, or adults in childbearing period not using an effective contraception method
* Treatment with any known non-marketed drug substance or experimental therapy within the longer of 5 terminal half-lives or 4 weeks prior to enrollment or currently participating in any other interventional clinical study
* Chronic or current infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment within two weeks prior to first study drug dose
* History of significant cerebrovascular disease in the past 6 months or ongoing event with active symptoms or sequelae
* HIV positive
* Significant concurrent, uncontrolled medical condition which may represent a risk for the patient
* Positive serology for HBV
* Positive serology for HCV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2014-11-11 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01-14 (Actual)

PRIMARY OUTCOMES:
Recommended dose | Day 21 of cycle 1 (3 weeks after start of treatment)
  During phase I, defined as the maximum Tolerable Dose of the BV in combination with ESHAP in relapsed/resistant HL patients.
Global response rate prior to ASCT | 9 weeks (after start of treatment)
  During phase II, Global response rate after BV-ESHAP as salvage regimen prior to ASCT.
Complete response | 9 weeks (after start of treatment)
  Percentage of patients with complete response rate after BV-ESHAP as salvage regimen prior to ASCT.

SECONDARY OUTCOMES:
Toxicity according to the CTC criteria | Prior every cycle, 14th day of first three cycles, at week 12, 16, 19, 22, 25, 31. Every 12 weeks for 2 years and then every 24 week up to 5 years.
  To determine the toxicity of BV-ESHAP regimen
Stem cell mobilization capacity | After first or second cycle of treatment
  To assess the stem cell mobilization capacity of the BV-ESHAP regimen: determine the expanse and effectiveness of the extraction of stem cells from peripheral blood.
Transplant-related mortality (TRM) | Prior every cycle, 14th day of first three cycles, at week 12, 16, 19, 22, 25, 31. Every 12 weeks for 2 years and then every 24 week up to 5 years.
Overall Survival (OS) | Prior every cycle, 14th day of first three cycles, at week 12, 16, 19, 22, 25, 31. Every 12 weeks for 2 years and then every 24 week up to 5 years.
  Percentage of patients alive after first dose of treatment through follow-up
Progression free survival (PFS) | Prior every cycle, 14th day of first three cycles, at week 12, 16, 19, 22, 25, 31. Every 12 weeks for 2 years and then every 24 week up to 5 years.
  Percentage of patients without progression of disease
Event-Free Survival | Prior every cycle, 14th day of first three cycles, at week 12, 16, 19, 22, 25, 31. Every 12 weeks for 2 years and then every 24 week up to 5 years.
  Percentage of patients without event
Time to HL Progression | Prior every cycle, 14th day of first three cycles, at week 12, 16, 19, 22, 25, 31. Every 12 weeks for 2 years and then every 24 week up to 5 years.
Disease-Free Survival | Prior every cycle, 14th day of first three cycles, at week 12, 16, 19, 22, 25, 31. Every 12 weeks for 2 years and then every 24 week up to 5 years.
Response Duration | Prior every cycle, 14th day of first three cycles, at week 12, 16, 19, 22, 25, 31. Every 12 weeks for 2 years and then every 24 week up to 5 years.
  Length of time between date of evidenced response and progression of disease or death
Lymphoma-Specific Survival | Prior every cycle, 14th day of first three cycles, at week 12, 16, 19, 22, 25, 31. Every 12 weeks for 2 years and then every 24 week up to 5 years.
Time to Next Treatment | Prior every cycle, 14th day of first three cycles, at week 12, 16, 19, 22, 25, 31. Every 12 weeks for 2 years and then every 24 week up to 5 years.

CONTACTS AND LOCATIONS:
Overall Officials: Ramón García-Sanz, MD, Study Chair — University of Salamanca
Locations (14):
- Spain (14):
  - Hospital Son Espases, Palma, Balearic Islands
  - Institut Català d'Oncologia, Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Institut Català d'Oncologia, Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital del Mar, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Clínico de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No